CLINICAL TRIAL: NCT01995032
Title: "A Double Blind Randomised Placebo Controlled Efficacy and Safety Study of L-citrulline and Metformin in Ambulant Children Aged Between 7 and 10 Years With Duchenne's Muscular Dystrophy"
Brief Title: L-citrulline and Metformin in Duchenne's Muscular Dystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMD02
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Duchenne's Muscular Dystrophy (DMD)
Keywords: Duchenne's muscular dystrophy; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 750 mg metformin and 7.5 g L-citrulline daily p.o. (Experimental): 7.5 g L-citrulline p.o. and 750 mg metformin daily p.o. (3x 2.5 g, respectively 3x 250 mg) for 26 weeks
  Interventions: Drug: 750 mg metformin and 7.5 g L-citrulline daily p.o.
- Placebo (Placebo Comparator): metformin placebo and L-citrulline placebo 3 times daily p.o. for 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 750 mg metformin and 7.5 g L-citrulline daily p.o.
  Arms: 750 mg metformin and 7.5 g L-citrulline daily p.o.
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to show that the intake of L-citrulline and metformin improves muscle function and delay of progression in patients with Duchenne's muscular dystrophy.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo controlled study. The study medication consists of L-citrulline and metformin, respectively placebo given orally; 2.5 g L-citrulline or placebo will be given 3 times daily, metformin containing 250 mg or placebo will be administered 3 times daily. The duration of the study is 26 weeks and comprehends one screening and three study visits.

Amendment 1: Amended eligibility criteria

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of DMD
* Patients 6.5 - 10 years of age at time of screening
* Ambulant
* Ability to walk 150 m in the 6 min walking distance (6MWT)
* D1 subdomain of the MFM scale >40%
* stable treatment with steroids for >6 months or steroid naïve patients

Exclusion Criteria:

* Previous (3 months or less) or concomitant participation in another therapeutic trial
* Use of L-citrulline, L-arginine or metformin within the last 3 months
* Known individual hypersensitivity to L-citrulline or metformin
* known or suspected malignancy
* Other chronic disease or clinical relevant limitation of renal, liver, heart function according to discretion of investigator
* start of cortisone treatment or change in dosage <6 months prior to screening

Ages: 78 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Mean change of motor function measure (MFM) D1 subscore (assessing standing and transfers) | baseline to week 26

SECONDARY OUTCOMES:
Mean change of MFM total score, the D2, and D3 MFM subscores | baseline to week 26
Mean change of six minute walking distance (6MWD) | baseline to week 26
Change of quantitative muscle MRI (Magnetic Resonance Imaging) including muscle fat content (MFC) and T2 times of thigh muscles | baseline to week 26
Change in the plasma/urine concentration for markers of muscle necrosis, oxidative stress, nitrosative stress, and change of microRNA (miRNA) | baseline to week 26
Mean change of quantitative muscle force (QMT) of knee extension and elbow flexion using hand held dynamometry (HHD) | baseline to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — University Children's Hospital Basel
Locations (1):
- University Children's Hospital, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Hafner P, Bonati U, Klein A, Rubino D, Gocheva V, Schmidt S, Schroeder J, Bernert G, Laugel V, Steinlin M, Capone A, Gloor M, Bieri O, Hemkens LG, Speich B, Zumbrunn T, Gueven N, Fischer D. Effect of Combination l-Citrulline and Metformin Treatment on Motor Function in Patients With Duchenne Muscular Dystrophy: A Randomized Clinical Trial. JAMA Netw Open. 2019 Oct 2;2(10):e1914171. doi: 10.1001/jamanetworkopen.2019.14171. PMID 31664444
- [Derived] Hafner P, Bonati U, Rubino D, Gocheva V, Zumbrunn T, Gueven N, Fischer D. Treatment with L-citrulline and metformin in Duchenne muscular dystrophy: study protocol for a single-centre, randomised, placebo-controlled trial. Trials. 2016 Aug 3;17(1):389. doi: 10.1186/s13063-016-1503-1. PMID 27488051